CLINICAL TRIAL: NCT00485797
Title: Effects of Methylphenidate on Postural Stability of Children Suffer From Attention Deficit Hyperactivity Disorder (ADHD) Under Single and Dual Task Conditions.
Brief Title: Effects of Ritalin on Postural Stability of Hyper Active Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Itshak Melzer PhD, PT, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR454707CTIL; MZ4547
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2007-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: attention deficit hyperactivity disorder (ADHD); Dual tasking; Postural Control; Methylphenidate (Ritalin); The focus of the study is To explore the effects of Ritalin on postural control in ADHD Children, during single and dual task conditions.
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ritalin — The effect of ritalin on postural stability of ADHD childrens will be measured using RCT study design

SUMMARY:
Experimental design overview The proposed project is a prospective experimental study design. Children (age <15) suffer from attention deficit hyperactivity disorder (ADHD) that their Parents willing to participate in the study will be tested with well-established measuring techniques of Balance control before and 1 hour after taking of Methylphenidate (Ritalin) in the movement and Rehabilitation Laboratory at BGU. An automated algorithm will be used to extract standardized stabilogram-diffusion parameters from each of the COP data sets collected during quiet standing. These parameters include diffusion coefficients, critical displacement, critical time and scaling exponents for both lateral and anterior-posterior sway directions (Collins & De Luca, 1993). For each of the conditions (before and 1 hour after the use of Ritalin) in three task conditions single task; dual task (concentrating and identifying specific music); and just Listening to a relaxing music. Participants will be required to stand on the platform 10 times for 30 s. For each trial, they will be instructed to sway as little as possible.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years old
* Diagnosed as ADHD childrens by a neurologist
* Taking methylphenidate (Ritalin)

Exclusion Criteria:

* Children who suffer from CP, or other neurological disease
* Children who suffer from psychiatric state
* Children who suffer from orthopedic condition (1/2 a year after a fracture in the lower limb)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Postural sway measures | Time 1: pre test' and hour later time 2: post testinng proceedure

CONTACTS AND LOCATIONS:
Overall Officials: Itshak Melzer, Dr, Principal Investigator — Ben-gurion University of the Negev, Beer-Sheva, Israel; Zmir Shorer, Dr, Study Chair — Soroka Medical Centar; Press Yossi, Prof, Study Director — Soroka University Medical Center
Locations (1):
- SorokaUMC, Beersheba, Israel